CLINICAL TRIAL: NCT04508309
Title: Phase 3 Randomized, Active-Comparator Controlled, Open-Label Trial to Evaluate the Immunogenicity & Safety of Alternate 2-Dose Regimens of Cecolin® Compared to Gardasil® in 9-14 Year-Old Girls in Low and Low-Middle Income Countries
Brief Title: Phase 3 Trial of a Bivalent Human Papilloma Virus (HPV) Vaccine (Cecolin®) in Young Girls
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Malaria Research Centre, Agogo Presbyterian Hospital, Ghana (Unknown); Frederick National Laboratory for Cancer Research, Leidos Biomedical Research, Inc., USA (Unknown); The Emmes Company, LLC (Industry); Xiamen Innovax Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CVIA-087
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cecolin® at 0 and 6 months (Experimental): Two doses of Cecolin® given at 0 and 6 months with blood draw at baseline, prior to second dose, one-month post second dose and 24 months after first dose
  Interventions: Biological: Cecolin®
- Cecolin® at 0 and 12 months (Experimental): Two doses of Cecolin® given at 0 and 12 months with blood draw at baseline, prior to second dose and one-month post second dose
  Interventions: Biological: Cecolin®
- Cecolin® at 0 and 24 months (Experimental): Two doses of Cecolin® given at 0 and 24 months with blood draw at baseline, prior to second dose and one-month post second dose
  Interventions: Biological: Cecolin®
- Gardasil® at 0 and 6 months (Active Comparator): Two doses of Gardasil® given at 0 and 6 months with blood draw at baseline, prior to second dose, one-month post second dose and 24 months after first dose
  Interventions: Biological: Gardasil®
- Gardasil® at 0 and Cecolin® at 24 months (Other): One dose of Gardasil® at 0 months and one dose of Cecolin® at 24 months with blood draw at baseline, prior to second dose and one-month post second dose.
  Interventions: Biological: Cecolin®; Biological: Gardasil®

INTERVENTIONS:
Biological: Cecolin® — Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine
  Arms: Cecolin® at 0 and 12 months; Cecolin® at 0 and 24 months; Cecolin® at 0 and 6 months; Gardasil® at 0 and Cecolin® at 24 months
Biological: Gardasil® — Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine
  Arms: Gardasil® at 0 and 6 months; Gardasil® at 0 and Cecolin® at 24 months

SUMMARY:
This randomized controlled trial will evaluate a bivalent HPV vaccine, Cecolin®, in alternate 2-dose regimens, compared to an established HPV vaccine. Gardasil® will be used as the comparator vaccine, as this vaccine is most widely used in low- and low-middle income countries.

DETAILED DESCRIPTION:
This randomized, active-comparator controlled, open-label study will enroll total of approximately 1025 girls aged 9 to 14 years, in one country in Africa (Ghana) and one country in South/Southeast Asia (Bangladesh). Participants will be randomized 1:1:1:1:1 to receive Cecolin® at 0 and 6 months, 0 and 12 months, or 0 and 24 months, Gardasil® at 0 and 6 months, or Gardasil® at 0 months and Cecolin® at 24 months. For each arm, blood will be collected for immunologic testing at baseline and one month following second dose. Additional blood collections will occur immediately prior to the administration of the second dose, as well as at additional later time points, for immunobridging to other published and ongoing trials. The study also aims to evaluate the performance of a mixed arm (group 5) of Gardasil® followed by Cecolin® and collect data on effects of interchangeability.

Girls of target age will be identified, and their parents contacted to attend an informational session for individual discussion, informed consent, assent and randomization.

The study will be conducted by the research groups in International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b) in Bangladesh and the Malaria Research Center (MRC) in Ghana.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (determined by investigator's assessment following medical history and physical examination, laboratory evaluation could be performed at the investigator's discretion) female between the ages of 9 - 14 years (all inclusive) at time of enrollment
2. Ability and willingness to provide parental consent and, if applicable based on local in-country regulations, participant assent
3. Parent/Legally Acceptable Representative provides informed consent
4. Anticipated ability and willingness to complete all study visits and evaluations
5. Living within the catchment area of the study without plans to move during the conduct of the study

Exclusion Criteria:

1. Presence of fever or acute disease on the day of vaccination (oral or axillary temperature ≥ 38˚ C)
2. If participants have childbearing potential, must not be breastfeeding or confirmed pregnant
3. Receipt of an investigational product within 30 days prior to randomization
4. Receipt of blood and/or blood products (including immunoglobulin) 3 months prior to any dose of vaccination or blood sampling
5. Receipt of a live virus vaccine (varicella virus containing vaccine, any measles, mumps, or rubella virus containing vaccine such as Measles, Mumps, and Rubella (MMR), or yellow fever vaccine but not including live attenuated influenza virus vaccine) 4 weeks prior and after each dose of HPV vaccine
6. History of any physical, mental, or developmental disorder that may hinder a participant's ability to comply with the study requirements
7. Any malignancy or confirmed or suspected immunodeficient condition such as HIV infection, based on medical history and physical examination
8. Receipt of or history of receipt of any medications or treatments that affect the immune system
9. Allergies to any components of the vaccine
10. Current or former participation in HPV vaccine related research.
11. Prior receipt of an investigational or licensed HPV vaccine
12. Any other condition(s) that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the participant unable to comply with the protocol

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 1025 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh
- Malaria Research Centre, Agogo Presbyterian Hospital, Agogo, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zaman K, Schuind AE, Adjei S, Antony K, Aponte JJ, Buabeng PB, Qadri F, Kemp TJ, Hossain L, Pinto LA, Sukraw K, Bhat N, Agbenyega T. Safety and immunogenicity of Innovax bivalent human papillomavirus vaccine in girls 9-14 years of age: Interim analysis from a phase 3 clinical trial. Vaccine. 2024 Apr 2;42(9):2290-2298. doi: 10.1016/j.vaccine.2024.02.077. Epub 2024 Mar 1. PMID 38431444
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Agbenyega T, Schuind AE, Adjei S, Antony K, Aponte JJ, Buabeng PBY, Clemens JD, Hossain L, Kemp TJ, Mercer LD, Pinto LA, Qadri F, Sukraw K, Bhat N, Zaman K. Immunogenicity and safety of an Escherichia coli-produced bivalent human papillomavirus vaccine (Cecolin) in girls aged 9-14 years in Ghana and Bangladesh: a randomised, controlled, open-label, non-inferiority, phase 3 trial. Lancet Infect Dis. 2025 Aug;25(8):861-872. doi: 10.1016/S1473-3099(25)00031-3. Epub 2025 Mar 19. PMID 40120597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in one clinical site in Bangladesh and one clinical site in Ghana.
Pre-assignment Details: Participants were randomized approximately equally within site into one of five treatment groups.
Groups:
- 1. Cecolin at Month 0 and 6: Participants received two doses of Cecolin 6 months apart (at Month 0 and Month 6).
- 2. Cecolin at Month 0 and 12: Participants received two doses of Cecolin 12 months apart (at Month 0 and Month 12).
- 3. Cecolin at Month 0 and 24: Participants received two doses of Cecolin 24 months apart (at Month 0 and Month 24).
- 4. Gardasil at Month 0 and 6: Participants received two doses of Gardasil 6 months apart (at Month 0 and Month 6)
- 5. Gardasil at Month 0 and Cecolin at Month 24: Participants received one dose of Gardasil at Month 0 and one dose of Cecolin at Month 24.
Period: Overall Study
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Started | 205 | 206 | 204 | 205 | 205
Received First Vaccination | 205 | 206 | 204 | 205 | 205
Received Second Vaccination | 205 | 204 | 199 | 205 | 201
Completed | 205 | 206 | 203 | 204 | 203
Not Completed | 0 | 0 | 1 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24 | Total
Number analyzed (Participants) | 205 | 206 | 204 | 205 | 205 | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (1.46) | 11.4 (1.37) | 11.4 (1.47) | 11.3 (1.39) | 11.3 (1.49) | 11.3 (1.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 206 | 204 | 205 | 205 | 1025
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 135 | 136 | 134 | 135 | 135 | 675
  Black | 70 | 70 | 70 | 70 | 70 | 350
Region of Enrollment [Number; unit: participants]
  Ghana | 70 | 70 | 70 | 70 | 70 | 350
  Bangladesh | 135 | 136 | 134 | 135 | 135 | 675

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) of Anti-HPV-16 Immunoglobulin G (IgG) Antibodies One Month After the Second Dose
Description: Anti-HPV-16 IgG antibodies were measured using HPV-16 virus-like particle (VLP) enzyme-linked immunosorbent assay (ELISA) one month after the second dose at the Frederick National Laboratory for Cancer Research in Frederick, Maryland, United States. The lower limit of quantitation of the HPV-16 assay was 1.41 international units (IU)/mL.
Time Frame: One month after the second dose (Month 7 for Groups 1 & 4, Month 13 for Group 2, and Month 25 for Groups 3 & 5).
Population: The Per Protocol Population includes participants who had no major protocol deviations that were determined to potentially interfere with the immunogenicity assessment of the study vaccine, were HPV-16 antibody negative at baseline, and had a valid serology result one month after second dose.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 198 | 189 | 190 | 194 | 193
IU/mL | 1507.4 [1329.0 to 1709.7] | 2408.7 [2116.0 to 2741.8] | 3326.1 [2960.6 to 3736.7] | 1352.4 [1199.1 to 1525.3] | 2387.3 [2091.4 to 2725.1]
Statistical Analysis 1: Comparison: 1. Cecolin at Month 0 and 6 vs 4. Gardasil at Month 0 and 6; The primary objective included three non-inferiority comparisons of Cecolin at 0 and 6 months, 0 and 12 months, or 0 and 24 months compared to Gardasil at 0 and 6 months. To control the type I error for the three co-primary non-inferiority hypotheses, a Bonferroni correction corresponding to 98.3% confidence intervals (CI) was used; Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower bound of the 98.3% confidence interval of the geometric mean concentration (GMC) ratio was greater than the non-inferiority margin of 0.5 for both HPV-16 and HPV-18; GMC Ratio = 1.09, 98.3% CI 2-sided [0.891 to 1.327] — GMC ratios (Cecolin/Gardasil) and corresponding confidence limits were calculated using linear models of the log concentration values adjusted by site and transformed back to the original scale
Statistical Analysis 2: Comparison: 2. Cecolin at Month 0 and 12 vs 4. Gardasil at Month 0 and 6; The primary objective included three non-inferiority comparisons of Cecolin at 0 and 6 months, 0 and 12 months, or 0 and 24 months compared to Gardasil at 0 and 6 months. To control the type I error for the three co-primary non-inferiority hypotheses, a Bonferroni correction corresponding to 98.3% CI was used; Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower bound of the 98.3% confidence interval of the GMC ratio was greater than the non-inferiority margin of 0.5 for both HPV-16 and HPV-18; GMC Ratio = 1.78, 98.3% CI 2-sided [1.455 to 2.176] — GMC ratio (Cecolin/Gardasil) and corresponding confidence limits were calculated using linear models of the log concentration values adjusted by site and transformed back to the original scale
Statistical Analysis 3: Comparison: 3. Cecolin at Month 0 and 24 vs 4. Gardasil at Month 0 and 6; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMC Ratio = 2.37, 98.3% CI 2-sided [1.942 to 2.903] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Geometric Mean Concentration of Anti-HPV-18 Immunoglobulin G Antibodies One Month After the Second Dose
Description: Anti-HPV-18 IgG antibodies were measured using HPV-18 VLP ELISA one month after the second dose at the Frederick National Laboratory for Cancer Research in Frederick, Maryland, United States. The lower limit of quantitation of the HPV-18 assay was 1.05 IU/mL.
Time Frame: One month after the second dose (Month 7 for Groups 1 & 4, Month 13 for Group 2, and Month 25 for Groups 3 & 5).
Population: The Per Protocol Population includes participants who had no major protocol deviations that were determined to potentially interfere with the immunogenicity assessment of the study vaccine, were HPV-18 antibody negative at baseline, and had a valid serology result one month after second dose.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 200 | 198 | 191 | 197 | 192
IU/mL | 382.7 [337.8 to 433.6] | 534.7 [469.4 to 609.1] | 535.2 [474.9 to 603.3] | 306.1 [269.3 to 347.9] | 379.0 [327.7 to 438.3]
Statistical Analysis 1: Comparison: 1. Cecolin at Month 0 and 6 vs 4. Gardasil at Month 0 and 6; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMC Ratio = 1.25, 98.3% CI 2-sided [1.022 to 1.539] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2. Cecolin at Month 0 and 12 vs 4. Gardasil at Month 0 and 6; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMC Ratio = 1.68, 98.3% CI 2-sided [1.372 to 2.069] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 3. Cecolin at Month 0 and 24 vs 4. Gardasil at Month 0 and 6; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMC Ratio = 1.71, 98.3% CI 2-sided [1.389 to 2.102] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-HPV-16 Neutralizing Antibodies
Description: Anti-HPV 16 serum neutralizing antibodies were measured in a subset of participants by pseudovirion-based neutralization assay (PBNA) at the Frederick National Laboratory for Cancer Research in Frederick, Maryland, United States. The lower limit of quantitation of the HPV-16 PBNA was a titer of < 21.
  Samples were collected prior to the second dose and 1 month after the second dose for all treatment groups, and 18 months after the second dose for participants in Groups 1 and 4.
Time Frame: Prior to 2nd dose (Month 6 for Groups 1 & 4, Month 12 for Group 2, and Month 24 for Groups 3 & 5), one month post 2nd dose (Month 7 for Groups 1 & 4, Month 13 for Group 2, and Month 25 for Groups 3 & 5) and 18 months after 2nd dose for Groups 1 and 4 only
Population: Per Protocol Population, PBNA Subset
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 40 | 41 | 41 | 40 | 40
titer
  Prior to Second Dose | 104.0 [78.6 to 137.7] | 95.1 [73.3 to 123.4] | 125.7 [95.3 to 165.6] | 71.6 [53.5 to 95.9] | 125.4 [85.2 to 184.5]
  One Month after Second Dose: number analyzed (Participants) | 40 | 41 | 40 | 40 | 38
  One Month after Second Dose | 16790.9 [11641.2 to 24218.6] | 32019.5 [25010.5 to 40992.7] | 48615.4 [36061.1 to 65540.5] | 14281.3 [10531.8 to 19365.7] | 31459.0 [24294.7 to 40736.0]
  18-Months after Second Dose: number analyzed (Participants) | 40 | 0 | 0 | 40 | 0
  18-Months after Second Dose | 1541.9 [1076.9 to 2207.5] |  |  | 1368.1 [998.8 to 1874.0] |

4. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-HPV-18 Neutralizing Antibodies
Description: Anti-HPV 18 serum neutralizing antibodies were measured in a subset of participants by pseudovirion-based neutralization assay (PBNA) at the Frederick National Laboratory for Cancer Research in Frederick, Maryland, United States. The lower limit of quantitation of the HPV-18 PBNA was a titer of < 16.
  Samples were collected prior to the second dose and 1 month after the second dose for all treatment groups, and 18 months after the second dose for participants in Groups 1 and 4.
Time Frame: as for outcome 3
Population: Per Protocol Population, PBNA Subset
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 40 | 41 | 40 | 41 | 41
titer
  Prior to Second Dose | 65.9 [42.1 to 103.2] | 51.1 [40.7 to 64.2] | 77.9 [58.1 to 104.5] | 47.6 [38.9 to 58.2] | 55.8 [36.3 to 85.6]
  One Month after Second Dose: number analyzed (Participants) | 40 | 41 | 39 | 41 | 39
  One Month after Second Dose | 6081.5 [3547.7 to 10425.1] | 9303.8 [7111.0 to 12172.7] | 11205.3 [8351.2 to 15034.8] | 6774.4 [5044.5 to 9097.6] | 7548.9 [5473.5 to 10411.2]
  18-Months after Second Dose: number analyzed (Participants) | 40 | 0 | 0 | 41 | 0
  18-Months after Second Dose | 441.7 [301.8 to 646.5] |  |  | 423.4 [289.8 to 618.5] |

5. Secondary Outcome: Seroconversion Rate For HPV-16 One Month After the Second Dose
Description: Seroconversion rate is defined as the percentage of participants with a 4-fold rise in anti-HPV 16 IgG antibodies as measured by ELISA from baseline one month following the second dose.
Time Frame: Baseline and one month after second dose (Month 7 for Groups 1 & 4, Month 13 for Group 2, and Month 25 for Groups 3 & 5).
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 198 | 189 | 190 | 194 | 193
percentage of participants | 100 | 100 | 100 | 100 | 100

6. Secondary Outcome: Seroconversion Rate For HPV-18 One Month After the Second Dose
Description: Seroconversion rate is defined as the percentage of participants with a 4-fold rise from baseline in anti HPV-18 IgG antibodies as measured by ELISA one month following the second dose.
Time Frame: as for outcome 5
Population: Per Protocol Population
Measure: Number; unit: percentage of participants
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 200 | 198 | 191 | 197 | 192
percentage of participants | 100 | 100 | 100 | 100 | 100

7. Secondary Outcome: GMC of Anti-HPV-16 IgG Antibodies One Month After the Second Dose: Comparison of Gardasil/Cecolin Mixed Dose With Gardasil 2-dose Regimen
Description: Anti-HPV-16 IgG antibodies were measured using HPV-16 VLP ELISA one month after the second dose at the Frederick National Laboratory for Cancer Research in Frederick, Maryland, United States. The lower limit of quantitation of the HPV-16 assay was 1.41 IU/mL.
  Anti-HPV-16 IgG GMCs measured 1 month after the second dose were compared between the Gardasil at Month 0 and Cecolin at 24 months two-dose regimen (Group 5) and the Gardasil at Month 0 and 6 two-dose regimen (Group 4).
Time Frame: One month after the second dose (Month 7 for Group 4 and Month 25 for Group 5).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 194 | 193
IU/mL | 1352.4 [1199.1 to 1525.3] | 2387.3 [2091.4 to 2725.1]
Statistical Analysis 1: Comparison: 4. Gardasil at Month 0 and 6 vs 5. Gardasil at Month 0 and Cecolin at Month 24; Test type: Non-Inferiority — Non-inferiority of the Cecolin containing arm (Group 5) compared to Gardasil at months 0 and 6 (Group 4) was to be demonstrated if the lower limit of the 95% CI of the GMC ratio was greater than the non-inferiority margin of 0.5 for both HPV-16 and HPV-18; GMC Ratio = 1.75, 95% CI 2-sided [1.476 to 2.071] — GMC ratio (Cecolin containing arm (Group 5)/Gardasil (Group 4)) and corresponding confidence limits were calculated using linear models of the log concentration values adjusted by site and transformed back to the original scale

8. Secondary Outcome: GMC of Anti-HPV-18 IgG Antibodies One Month After the Second Dose: Comparison of Gardasil/Cecolin Mixed Dose With Gardasil 2-dose Regimen
Description: Anti-HPV-18 IgG antibodies were measured using HPV-18 VLP ELISA one month after the second dose at the Frederick National Laboratory for Cancer Research in Frederick, Maryland, United States. The lower limit of quantitation of the HPV-18 assay was 1.405 IU/mL.
  Anti-HPV-18 IgG GMCs measured 1 month after the second dose were compared between the Gardasil at Month 0 and Cecolin at 24 Months two-dose regimen (Group 5) and the Gardasil at Month 0 and 6 two-dose regimen (Group 4).
Time Frame: One month after the second dose (Month 7 for Group 4 and Month 25 for Group 5).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 197 | 192
IU/mL | 306.1 [269.3 to 347.9] | 379.0 [327.7 to 438.3]
Statistical Analysis 1: Comparison: 4. Gardasil at Month 0 and 6 vs 5. Gardasil at Month 0 and Cecolin at Month 24; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; GMC Ratio = 1.21, 95% CI 2-sided [1.004 to 1.451] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: GMC of Anti-HPV-16 IgG Antibodies 18-Months After Second Dose
Description: Anti-HPV-16 IgG antibodies were measured using HPV-16 VLP ELISA 18 months after the second dose for participants who received a 6-month dosing regimen (Groups 1 and 4) only.
Time Frame: 18 months after the second dose (Month 24)
Population: The Per Protocol Population includes participants who had no major protocol deviations that were determined to potentially interfere with the immunogenicity assessment of the study vaccine, were HPV-16 antibody negative at baseline, and had a valid serology result 18-months after the second dose. Only participants who received the 6 month dose regimens were assessed for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 1. Cecolin at Month 0 and 6 | 4. Gardasil at Month 0 and 6
Number analyzed (Participants) | 198 | 195
IU/mL | 138.5 [120.8 to 158.7] | 119.1 [104.1 to 136.2]
Statistical Analysis 1: Comparison: 1. Cecolin at Month 0 and 6 vs 4. Gardasil at Month 0 and 6; Test type: Non-Inferiority — Non-inferiority of Cecolin at Months 0 and 6 (Group 1) compared to Gardasil at Months 0 and 6 (Group 4) was to be demonstrated if the lower limit of the 95% CI of the GMC ratio was greater than the non-inferiority margin of 0.5 for both HPV-16 and HPV-18; GMC Ratio = 1.12, 95% CI 2-sided [0.933 to 1.344] — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: GMC of Anti-HPV-18 IgG Antibodies 18-Months After Second Dose
Description: Anti-HPV-18 IgG antibodies were measured using HPV-18 VLP ELISA 18 months after the second dose for participants who received a 6-month dosing regimen (Groups 1 and 4) only.
Time Frame: 18 months after the second dose (Month 24)
Population: The Per Protocol Population includes participants who had no major protocol deviations that were determined to potentially interfere with the immunogenicity assessment of the study vaccine, were HPV-18 antibody negative at baseline, and had a valid serology result 18 months after the second dose. Only participants who received the 6-month dosing regimens were assessed for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 1. Cecolin at Month 0 and 6 | 4. Gardasil at Month 0 and 6
Number analyzed (Participants) | 200 | 198
IU/mL | 30.2 [25.9 to 35.2] | 23.2 [19.8 to 27.3]
Statistical Analysis 1: Comparison: 1. Cecolin at Month 0 and 6 vs 4. Gardasil at Month 0 and 6; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; GMC Ratio = 1.32, 95% CI 2-sided [1.070 to 1.635] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Participants With Solicited Adverse Events
Description: Solicited adverse events (AEs) were assessed by study staff 30 minutes after each vaccination and then daily for seven days after each vaccination by the participants using a memory aid.
  The following specific solicited AEs were monitored for this trial:
  * Local Reactions:
    * Pain, erythema/redness, swelling, induration, pruritus, abscess.
  * General/Systemic Reactions:
    * Fever (oral or axillary temperature ≥ 38.0°C), headache, vomiting, nausea, fatigue, chills, muscle pain, cough, diarrhea, dizziness, allergic dermatitis, rash, syncope, and anorexia.
Time Frame: For 30 minutes after each vaccination and for up to 7 days after each vaccination
Population: Total Vaccinated Population includes all randomized participants who received at least one dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 205 | 206 | 204 | 205 | 205
Participants
  Within 30 Minutes of Vaccination: Any Local Reactions | 4 | 15 | 2 | 12 | 5
  Within 30 Minutes of Vaccination: Any Systemic Reactions | 12 | 3 | 7 | 10 | 7
  Within 7 Days of Vaccination: Any Local Reactions | 131 | 113 | 106 | 138 | 120
  Within 7 Days of Vaccination: Any Systemic Reactions | 72 | 59 | 48 | 76 | 50

12. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Unsolicited AEs were any AEs reported spontaneously by the participant, identified during interview at study visits, observed by the study personnel during study visits or those identified during review of medical records or source documents. Unsolicited AEs were events occurring from the time of each study injection through approximately 30 days after each vaccination. Solicited AEs with onset after the solicitation period and through Day 30 post-vaccination were captured as unsolicited AEs.
Time Frame: For 30 days after each dose (Month 0 (all groups), Month 6 (Groups 1 and 4), Month 12 (Group 2), and Month 24 (Groups 3 and 5)
Population: Total Vaccinated Population includes all randomized participants who received at least one dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 205 | 206 | 204 | 205 | 205
Participants | 43 | 41 | 46 | 52 | 34

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was any AE that resulted in any of the following outcomes:
  1. Death
  2. Was life-threatening
  3. Required inpatient hospitalization or prolongation of existing hospitalization.
  4. Resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
  5. Congenital abnormality or birth defect.
  6. Important medical event that may not have resulted in one of the above outcomes but may have jeopardized the health of the study participant or (and) required medical or surgical intervention to prevent one of the outcomes listed in the above definition of SAEs.
  SAEs were collected from the time of first vaccination through the end of the study for each participant.
Time Frame: From first dose through the end of study (up to 730 days for Groups 1 and 4, 395 days for Group 2, and 760 days for Groups 3 and 5)
Population: Total Vaccinated Population includes all randomized participants who received at least one dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 205 | 206 | 204 | 205 | 205
Participants | 4 | 0 | 5 | 4 | 3

14. Other Pre Specified Outcome: GMC of Anti-HPV-16 IgG Antibodies Prior to the Second Dose
Description: To evaluate the persistence of antibody responses to HPV after a single dose of vaccine, anti-HPV-16 IgG antibodies were measured using HPV-16 VLP ELISA immediately prior to the second dose.
Time Frame: Prior to the second dose (Month 6 for Groups 1 & 4, Month 12 for Group 2, and Month 24 for Groups 3 & 5).
Population: The Per Protocol Population includes participants who had no major protocol deviations that were determined to potentially interfere with the immunogenicity assessment of the study vaccine, were HPV-16 antibody negative at baseline, and had a valid serology result prior to receiving the second dose.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 198 | 191 | 193 | 196 | 197
IU/mL | 17.5 [15.6 to 19.7] | 12.6 [11.0 to 14.6] | 12.0 [10.3 to 13.9] | 11.1 [9.9 to 12.3] | 10.5 [9.0 to 12.3]

15. Other Pre Specified Outcome: GMC of Anti-HPV-18 IgG Antibodies Prior to the Second Dose
Description: To evaluate the persistence of antibody responses to HPV after a single dose of vaccine, anti-HPV-18 IgG antibodies were measured using HPV-16 VLP ELISA immediately prior to the second dose.
Time Frame: Prior to the second dose (Month 6 for Groups 1 & 4, Month 12 for Group 2, and Month 24 for Groups 3 & 5).
Population: The Per Protocol Population includes participants who had no major protocol deviations that were determined to potentially interfere with the immunogenicity assessment of the study vaccine, were HPV-18 antibody negative at baseline, and had a valid serology result prior to receiving the second dose.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
Number analyzed (Participants) | 200 | 200 | 195 | 199 | 196
IU/mL | 6.5 [5.9 to 7.3] | 4.3 [3.8 to 4.9] | 4.4 [3.8 to 5.1] | 4.1 [3.6 to 4.6] | 3.2 [2.7 to 3.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the end of study; up to 730 days for Groups 1 and 4, 395 days for Group 2, and 760 days for Groups 3 and 5.
Arm/Group | 1. Cecolin at Month 0 and 6 | 2. Cecolin at Month 0 and 12 | 3. Cecolin at Month 0 and 24 | 4. Gardasil at Month 0 and 6 | 5. Gardasil at Month 0 and Cecolin at Month 24
All-Cause Mortality (participants affected / at risk) | 0/205 | 0/206 | 0/204 | 0/205 | 1/205
Serious Adverse Events (participants affected / at risk) | 4/205 | 0/206 | 5/204 | 4/205 | 3/205
Other Adverse Events (participants affected / at risk) | 155/205 | 145/206 | 130/204 | 165/205 | 145/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1. Cecolin at Month 0 and 6 (N=205) | 2. Cecolin at Month 0 and 12 (N=206) | 3. Cecolin at Month 0 and 24 (N=204) | 4. Gardasil at Month 0 and 6 (N=205) | 5. Gardasil at Month 0 and Cecolin at Month 24 (N=205)
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Typhoid fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1. Cecolin at Month 0 and 6 (N=205) | 2. Cecolin at Month 0 and 12 (N=206) | 3. Cecolin at Month 0 and 24 (N=204) | 4. Gardasil at Month 0 and 6 (N=205) | 5. Gardasil at Month 0 and Cecolin at Month 24 (N=205)
Nausea (Gastrointestinal disorders) | 8 | 6 | 7 | 6 | 5
Vomiting (Gastrointestinal disorders) | 6 | 2 | 5 | 10 | 2
Gastritis (Gastrointestinal disorders) | 5 | 5 | 4 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 3 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 5 | 7 | 1
Vaccination site pain (General disorders) | 133 | 119 | 106 | 141 | 121
Fatigue (General disorders) | 5 | 2 | 10 | 5 | 6
Pyrexia (General disorders) | 5 | 3 | 4 | 9 | 4
Chills (General disorders) | 6 | 3 | 2 | 9 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 10 | 10 | 10 | 11
Malaria (Infections and infestations) | 9 | 7 | 11 | 9 | 6
Urinary tract infection (Infections and infestations) | 6 | 8 | 5 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 6 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 6 | 7 | 22 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3 | 3 | 3
Headache (Nervous system disorders) | 40 | 36 | 33 | 50 | 31
Dizziness (Nervous system disorders) | 11 | 8 | 8 | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 14 | 5 | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT04508309/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT04508309/SAP_001.pdf